CLINICAL TRIAL: NCT06241807
Title: A Phase II Trial of Neoadjuvant Camrelizumab Combined With Chemotherapy for Resectable Stage IIIA-IIIB Non-Small Cell Lung Cancer
Brief Title: Neoadjuvant Camrelizumab Combined With Chemotherapy for Resectable Stage IIIA-IIIB NSCLC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shandong Cancer Hospital and Institute (Other)
Responsible Party: Principal Investigator, Xue Meng, MD, PhD, Shandong Cancer Hospital and Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SDZL-MX-01
Record Dates: First submitted 2024-01-28; First posted 2024-02-05 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: IMMUNOTHERAPY; Neoadjuvant Therapy; Resectable Lung Non-Small Cell Carcinoma; Biomarkers / Blood
Keywords: Camrelizumab; Non-Small Cell Lung Cancer; Neoadjuvant Therapy; Biomarkers Analysis
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — camrelizumab; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Camrelizumab Plus Chemotherapy Arm (Experimental): Patients were assigned to receive 3 cycles of camrelizumab (200 mg) plus chemotherapy (nab-paclitaxel, 130 mg/m2 or pemetrexed (for adenocarcinoma), 500mg/m2 plus platinum [cisplatin, 75 mg/m2; carboplatin, area under the curve, 5])
  Interventions: Drug: Camrelizumab Plus Chemotherapy

INTERVENTIONS:
Drug: Camrelizumab Plus Chemotherapy — Patients were assigned to receive 3 cycles of camrelizumab (200 mg) plus chemotherapy (nab-paclitaxel, 130 mg/m2 or pemetrexed (for adenocarcinoma), 500mg/m2 plus platinum [cisplatin, 75 mg/m2; carboplatin, area under the curve, 5])

SUMMARY:
This study aims to evaluate the efficacy and safety of neoadjuvant camrelizumab combined with chemotherapy in resectable stage IIIA and IIIB (T3-4N2) non-small cell lung cancer (NSCLC) patients. Inclusion criteria are: age 18-75, pathologically confirmed resectable stage IIIA-IIIB (T3-4N2) NSCLC, absence of EGFR, ALK, and ROS1 gene mutations, and Eastern Cooperative Oncology Group (ECOG) status 0-1. All patients receive three cycles of camrelizumab combined with platinum-based doublet chemotherapy, followed by curative surgery within 4-6 weeks after completion of chemotherapy. Patients undergo 18F-fluorodeoxyglucose (FDG) PET/CT scans in 1 week before treatment and 1 week before surgery, and peripheral blood samples are collected for biomarker analysis. The primary endpoints for follow-up are pathologic complete response (pCR) rate and major pathological response (MPR) rate, while secondary endpoints include safety and progression-free survival. Exploratory endpoints include molecular imaging research and biomarker analysis.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75
* Pathologically confirmed resectable stage IIIA-IIIB (T3-4N2) NSCLC
* Absence of EGFR, ALK, and ROS1 gene mutations
* Eastern Cooperative Oncology Group (ECOG) status 0-1
* Signed written informed consent prior to the implementation of any trial-related rocedures
* Adequate organ function, evidenced by laboratory results with no contraindications to chemotherapy: Absolute neutrophil count ≥ 1,500 х109/L, Thrombocytes ≥ 100 х 109/L, Hemoglobin ≥ 90 mg/L, Creatinine ≤ 1.5 x ULN or creatinine clearance (calculated using the Cockcroft-Gault formula) ≥ 40 mL/min, Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) > 2.5 x upper limit of normal (ULN), Alkaline phosphatase (ALP) > 5 x ULN, Bilirubin > 1.5 х ULN

Exclusion Criteria:

* Patients diagnosed with any other malignant tumor
* Have received prior therapy with chemotherapy or immune checkpoint inhibitor
* Insufficient caloric and/or fluid intake despite consultation with a dietitian and/or tube feeding
* Have an active infection requiring systemic therapy that has not resolved 3 days (simple infection, such as cystitis) to 7 days (severe infection, such as pyelonephritis) before the first dose of trial treatment
* Patients who cannot tolerate chemoradiotherapy or surgery due to severe cardiac, lung dysfunction
* A history of interstitial lung disease or non-infectious pneumonia
* Active autoimmune disease with systemic therapy (ie, use of disease modifiers, corticosteroids, or immunosuppressive drugs) in the past 2 years
* Known history of human immunodeficiency virus (HIV) infection (i.e., positive for HIV 1/2 antibody) and various viral hepatitis infections
* Patients who have received allogeneic stem cell or solid organ transplantation
* Women during pregnancy or lactation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-12-02 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Major Pathological Response Rate | From date of surgery to 14 days later
  No more than 10% of tumor cells were found in neoadjuvant surgical specimens
Pathologic complete response rate | From date of surgery to 14 days later
  No histological evidence of malignancy was found in the primary tumor and metastatic lymph nodes

SECONDARY OUTCOMES:
Adverse events | 24 weeks
  Number and percentage of cases of all adverse events
Disease-free survival | 24 months
  The period of time from the initiation of treatment to the observation of disease progression or occurrence of death for any reason

OTHER OUTCOMES:
Molecular imaging research and biomarker analysis | 20 weeks
  Plasma ctDNA testing, serum metabolomics testing, 18F-FDG uptake value, circulating immunological biomarkers, and observation of tumor immune microenvironment

CONTACTS AND LOCATIONS:
Locations (1):
- Shandong Cancer Hospital and Institute, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wang K, Wang X, Meng X, Zhang G, Cai G. Molecular imaging using 18F-FDG PET/CT and circulating inflammatory and immune indicators to predict pathological response to neoadjuvant camrelizumab plus chemotherapy in resectable stage IIIA-IIIB NSCLC. Ann Nucl Med. 2025 Aug;39(8):862-874. doi: 10.1007/s12149-025-02057-0. Epub 2025 May 10. PMID 40348946